CLINICAL TRIAL: NCT04525729
Title: A Multicentre, Randomized, Controlled Study of Rituximab in Treatment of Primary IgA Nephropathy
Brief Title: Rituximab and RASi in Patients with IgAN
Acronym: RITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nan Chen,MD (Other)
Collaborators: Dongfang Hospital Affiliated to Tongji University (Other); Shanghai Pudong New Area People's Hospital (Other); Ruijin Hospital North Shanghai Jiao Tong University School of Medicine (Unknown); Ningbo Municipal Yinzhou District No.2 Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Xiamen Hong'ai Hospital (Unknown); Sir Run Run Shaw Hospital (Other); Tongji Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Nan Chen,MD, professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RITA
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: IgA Nephropathy
Keywords: IgAN; Rituximab; RASi; Gd-IgA1; proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Rituximab; resminostat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab+RASi(ACEI and/or ARB) (Experimental): The maximum tolerable dose of RASi will be using everyday depending on the individual factors of the subject, combined with rituximab 1g(D1, D31 respectively, intravenous infusion). Add 1 g rituximab at 6 months.
  Interventions: Drug: Rituximab; Drug: RAS 2410
- RASi(ACEI and/or ARB） (Other): The maximum tolerable dose of RASi will be using everyday depending on the individual factors of the subject.
  Interventions: Drug: RAS 2410

INTERVENTIONS:
Drug: Rituximab — To evaluate the efficacy and safety of HLX01 combined with RASi in patients with IgAN.
  Other Names: HLX01
  Arms: Rituximab+RASi(ACEI and/or ARB)
Drug: RAS 2410 — To evaluate the efficacy and safety of RASi in patients with IgAN.
  Other Names: No specific restrictions

SUMMARY:
A study to evaluate safety and activity in treatment of IgAN patients using Rituximab in combination with RASi(ACEI and/or ARB) compared with RASi.

DETAILED DESCRIPTION:
IgA nephropathy (IgAN, IgA nephropathy), is currently the most common glomerular disease worldwide, which is characterized by High population quantity, wide distribution, strong heterogeneity.

Diagnosis of Urinary protein control level within 1 year is one of the important predictors of renal failure in IgAN patients.Previous studies have shown that patients with renal insufficiency, hypertension, or urinary protein > 1g at 24h during renal biopsy, and those with poor urinary protein control within 1 year of follow-up, have a higher risk of disease progression, and more than 30-50% of patients will develop into end-stage renal disease (ESRD) within 10 years.

The recommended treatments for IgAN in the KDIGO guidelines include: RASi, glucocorticoid, immunosuppressor, antiplatelet drugs, lipid-lowering drugs, etc. Several trials have demonstrated the benefit of RASi in retarding disease progression in IgAN patients with proteinuria, but there is currently no specific treatment for IgAN.

In recent years, it has been found that excessive production of Galactos-deficient IgA1 is one of the initiating factors of the pathogenesis of IgAN. Infection by pathogenic microorganisms induces lymphocytes in IgAN patients to produce anti-GD-IgA1 autoantibodies (second strike), which forms circulating immune complexes to deposit in the kidney and activates complement, which is an important pathogenesis of IgAN.However, recent studies have suggested that B-cell depletion therapy is effective for many aabs mediated renal diseases (e.g., membranous nephropathy, lupus nephritis, etc.). Rituximab, which combined with CD20 antigen on the B cell surface, can deplete B cells and play a therapeutic role by reducing antibody production. Therefore, the treatment of rituximab has potential therapeutic value for IgAN patients as well.

However, there were very few studies which have shown the efficacy and safety of rituximab in the treatment of IgA nephropathy, only groups reported abroad, and the results were inconsistent. At present, there have been no randomized controlled studies to verify the safety and efficacy of rituximab in the treatment of IgA nephropathy, especially in Chinese with high incidence of IgAN.

In this study, treatment of rituximab combining with RASi will be compared with RASi for IgAN patients, to explore an effective and safer regimen for IgAN, so as to bring more hope to patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 to 75 of age, male or female;
* 2. primary IgA nephropathy confirmed by renal biopsy
* 3. eGFR>30ml/min/1.73m2(calculated according to the CKD-EPI formula);
* 4. After using maximum tolerated doses of ACEI and/or ARB for 3 months, the following two points should be met:

  1. 24h proteinuria ≥1g;
  2. Bp<130/80 mmHg；
* 5. Serum albumin > 25g/L;
* 6. Sign the informed consent.

Note : It is suggested that active IgAN patients should be selected. Active IgAN is specifically defined as conforming to any of the following :

1. ) intradermal augmentation ( E1 ),
2. ) crescentic body 0 - 50 % ( C1 / C2 ),
3. ) fibrinoid necrosis,
4. ) more interstitial inflammatory cell infiltration. At the same time, the proportion of sclerosis was low ( spherical or segmental sclerosis ball < 50 % ), and interstitial fibrosis was low ( below T2 ).

Exclusion Criteria:

* 1. Evidence of the use of glucocorticoids for immunosuppressive therapy, such as: nephrotic syndrome, pathology for small lesions with IgA nephropathy. or the proportion of crescents confirmed by renal biopsy within 12 months was more than 50 %.
* 2. Clinical confirmation of cirrhosis, chronic active liver disease, or hepatitis B, C, or HIV which can detect viral replication;
* 3. Clinically confirmed IgA nephropathy secondary to systemic diseases such as systemic lupus erythematosus, allergic purpura.
* 4. Patients with non-simple IgA nephropathy, such as diabetic nephropathy or obesity-related nephropathy.
* 5. A history of active systemic infection or severe infection occurred one month before enrollment.
* 6. Those who are pregnant or lactating or unwilling to take contraceptive measures.
* 7. Current or recent ( within 30 days ) exposure to any research drug.
* 8. Patients with allergic reactions to rituximab and / or known allergic reactions.
* 9. Laboratory tests meeting the following criteria should be excluded:

  (1) Hemoglobin <80g/L; (2) Platelet <80×10^9/L; (3) Neutrophils < 1.0×10^9/L; (4) Aspartic acid aminotransferase (AST) or alanine aminotransferase (ALT) >2.5× normal upper limit, except for the correlation with the primary disease;
* 10. Continuous use of hormones or other immunosuppressive therapy in the past 6 months;
* 11. Accompanying or past malignant tumors, except for fully treated skin basal or squamous cell carcinoma or cervical carcinoma in situ;
* 12. History of psychosis may interfere with normal participation in this study;
* 13. Patients with major heart or lung diseases (including obstructive pulmonary disease);
* 14. In acute and chronic tuberculosis infection period (tuberculin test positive, chest X-ray suspected tuberculosis patients);
* 15. Patients with history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* 16. Weight less than 50kg should be excluded;
* 17. Other researchers judge the patients unsuitable for inclusion in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in proteinuria levels over 1 year compared with baseline | 1 year
  Primary outcome included changes in proteinuria levels over 1 year compared with baseline

SECONDARY OUTCOMES:
The proportion of 50% reduction in mean urinary protein compared with baseline over 1 year | 1 year
  Statistical data of proportion of 50% reduction in mean urinary protein compared with baseline over 1 year
The proportion of 50% reduction in mean urinary protein compared with baseline over 6 months | 6 months
  Statistical data of proportion of 50% reduction in mean urinary protein compared with baseline over 6 months
Changes in proteinuria levels over 6 months compared with baseline | 6 months
  Secondary Outcome included changes in proteinuria levels over 6 months compared with baseline
Changes in eGFR levels over 1 year compared with baseline | 1 year
  To evaluate the efficacy of treatment in renal function
Changes in Gd-IgA1 levels | 1 year
  To observe the changes in GD-IGA1 level
Incidence of adverse events | 1 year
  Record the safety of Interventional drugs
Incidence of ESRD | 1 year
  Evaluate the efficacy of treatment
The proportion of 50% reduction in eGFR levels or doubling serum creatinine compared with baseline | 1 year
  To evaluate the renal function
Incidence of infection | 1 year
  To evaluate the safety of Rituximab

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xie, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639